CLINICAL TRIAL: NCT06555770
Title: Effects of Music and Stress Ball Application on Patients During Cataract Surgery Examining the Effect on Anxiety and Pain
Brief Title: Effects of Music and Stress Ball Application on Patients During Cataract Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Akdeniz University (Other)
Responsible Party: Principal Investigator, Seda Cansu Yeniğün, Lecturer Dr, Akdeniz University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2490Akdeniz
Record Dates: First submitted 2024-08-13; First posted 2024-08-15 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Cataract; Nursing Caries
Keywords: cataract; music intervention; stress ball; pain; anxiety
MeSH Terms: conditions — Cataract; Pain; Anxiety Disorders

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Stres topu grubu (Experimental): Pain levels will be tested with VAS 10 minutes before the surgery, and anxiety levels with the VAS-A and Spielberg Continuous Anxiety Scale. The stress balls will be given to both hands of the patient, counting to five and pressing twice. The patient will be shown to use the stress balls for 15 minutes during the surgery. The patient will be told to use the stress balls for 15 minutes during the surgery. After 15 minutes, the researcher will inform the patient and make sure the patient drops the balls.
  Interventions: Behavioral: müzik müdahalesi
- Müzik grubu (Experimental): Pain levels will be tested with VAS 10 minutes before the surgery, and anxiety levels with the VAS-A and Spielberg Continuous Anxiety Scale. According to the randomization, the patient in the music intervention group will first be asked by the researcher to select his favorite music from the playlist. The playlist will be created using the Spotify app. The playlist will include a total of 50 songs from each group (pop, Turkish art music, local Turkish and religious music), including ten songs. Options will be shown to the patient on the phone (Apple/MU783TU/A) and the music he wants will be added to the playlist.
  The patient will be told that the selected music will be listened to for 15 minutes during cataract surgery.
  Interventions: Behavioral: müzik müdahalesi
- Kontrol grubu (No Intervention): Pain levels will be tested with VAS 10 minutes before the surgery, and anxiety levels with the VAS-A and Spielberg Continuous Anxiety Scale. The patient in the control group will not be given any intervention.

INTERVENTIONS:
Behavioral: müzik müdahalesi — One group of patients will be listening to music for 15 minutes during the surgery, while the other group will be applied a stress ball.
  Other Names: stres topu
  Arms: Müzik grubu; Stres topu grubu

SUMMARY:
Cataract is one of the leading causes of preventable blindness in the world and in Türkiye. Cataract surgery is one of the most frequently performed and most reliable surgeries for eye diseases. Advances in anesthesia and surgical techniques make it possible for most cataract surgery procedures to be performed under topical anesthetic.

DETAILED DESCRIPTION:
This success greatly reduces the duration of surgery, and the side effects associated with local or general anesthesia. However, despite the sedation that can be administered before and during surgery (e.g. benzodiazepines and opioids), patients can experience significant anxiety along with a certain degree of pain and discomfort during surgery. Anxiety causes stress that causes the cardiovascular system to respond by activating the sympathetic nervous system, which causes an increase in heart rate and blood pressure (BP) levels. These mechanisms can complicate the surgical procedure due to increased intraocular pressure. Hypertension and tachycardia above 85 discharges per minute represent an increased risk of orbital bleeding during local anesthetic injection and potential perioperative supracoroidal expulsive bleeding. The sequence and pre-operative music intervention is to be an inexpensive, easy-to-implement technique that has no side effects, has no significant beneficial effects on the anxiety of patients in different surgical populations. Also, music intervention allows for better patient co-operation during surgery under topical anesthesia and a drop in intraoperative blood pressure. Another method that is effective in reducing anxiety and pain is the stress ball. The stress ball is usually a soft toy that is not greater than 7 cm, gets stuck, relieving stress and muscle tension, or manipulated with fingers for exercising the muscles. One of the methods of distracting attention, the stress ball is an effective way of ensuring cognitive focus. The stress ball method has been used to reduce patients' anxiety and pain. Stretching the stress ball during surgery increases the feeling of strength, allowing patients to have direct control over the object. In this way, surgical intervention has a positive effect on anxiety and patient satisfaction without intervention. While the literature includes studies involving the combination of stress ball use and music intervention on surgical patients, there is no research involving combined use of music and stress ball application in cataract surgery in a single study. The investigators work therefore contributes to literature.

ELIGIBILITY:
Inclusion Criteria:

* Being 18 years of age or older and undergoing PHACO surgery,
* Not having any hearing or perception problems,
* Not having any physical problems to squeeze a stress ball,
* Having undergone cataract surgery for the first time,
* Being willing to participate in the research.

Exclusion Criteria:

* Any use of any analgesic or anxiolytic within 24 hours prior to surgery,
* Transition from topical to general anesthesia during surgery,
* A psychiatric diagnosis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2024-08-20 (Actual); Primary Completion 2025-02-20 (Actual); Study Completion 2025-03-01 (Actual)

PRIMARY OUTCOMES:
Pain (Visual Analog Scale) | 15 minutes before surgery
  Grading is made with a 10 cm long horizontal or vertical ruler on the scale and "0" means no pain and "10" means the most severe pain.
  The patient marks the intensity of pain he feels on the ruler. If the marked value is between 1-4, it indicates mild pain, between 5-6 indicates moderate pain, and between 7-10 indicates severe pain.
  In the application, the patient was asked to mark the intensity of pain he felt on the ruler and the value was measured and recorded.
Pain (Visual Analog Scale) | During surgery
  Grading is made with a 10 cm long horizontal or vertical ruler on the scale and "0" means no pain and "10" means the most severe pain.
  The patient marks the intensity of pain he feels on the ruler. If the marked value is between 1-4, it indicates mild pain, between 5-6 indicates moderate pain, and between 7-10 indicates severe pain.
  In the application, the patient was asked to mark the intensity of pain he felt on the ruler and the value was measured and recorded.
Pain (Visual Analog Scale) | 10 minutes after surgery
  Grading is made with a 10 cm long horizontal or vertical ruler on the scale and "0" means no pain and "10" means the most severe pain.
  The patient marks the intensity of pain he feels on the ruler. If the marked value is between 1-4, it indicates mild pain, between 5-6 indicates moderate pain, and between 7-10 indicates severe pain.
  In the application, the patient was asked to mark the intensity of pain he felt on the ruler and the value was measured and recorded.
Anxiety (Visual Analog Scale-Anxiety) | 15 minutes before surgery
  Patients' anxiety will be evaluated (0-10 point). Grading is made with a 10 cm long horizontal or vertical ruler on the scale and "0" means no anxiety and "10" means the most severe anxiety.
  In the application, the patient was asked to mark the intensity of pain he felt on the ruler and the value was measured and recorded.
Anxiety (Visual Analog Scale-Anxiety) | During surgery
  Patients' anxiety will be evaluated (0-10 point). Grading is made with a 10 cm long horizontal or vertical ruler on the scale and "0" means no anxiety and "10" means the most severe anxiety.
  In the application, the patient was asked to mark the intensity of pain he felt on the ruler and the value was measured and recorded.
Anxiety (Visual Analog Scale-Anxiety) | 10 minutes after surgery
  Patients' anxiety will be evaluated (0-10 point). Grading is made with a 10 cm long horizontal or vertical ruler on the scale and "0" means no anxiety and "10" means the most severe anxiety.
  In the application, the patient was asked to mark the intensity of pain he felt on the ruler and the value was measured and recorded.
State-Trait Anxiety Inventory (STAI-II) | 15 minutes before surgery
  STAI-II is a well-researched clinical tool for evaluating the tendency towards anxiety. A cut-off point of 39-40 typically indicates clinically significant symptoms of a state of anxiety.

CONTACTS AND LOCATIONS:
Locations (1):
- Seda Cansu Yeniğün, Antalya, Kumluca, Turkey (Türkiye)